CLINICAL TRIAL: NCT02383446
Title: Evaluation of the Efficiency of Hydraulic Microprocessor Prosthetic Foot for Traumatic Transtibial Amputees
Brief Title: Efficiency of Hydraulic Microprocessor Prosthetic Foot for Traumatic Transtibial Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Itzhak Siev-Ner, Head of The Department of Orthopedic Rehabilitation, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-13-0292-SMC
Record Dates: First submitted 2015-02-25; First posted 2015-03-09 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Unilateral Transtibial Amputee
Keywords: Echeclon; Elan; TTA; Transtibial Amputee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elan foot prosthesis (Experimental): The research group will perform a gait analysis test (on a computerized treadmill) using their own non-computerized hydraulic foot, while in-socket pressures are measured. The prosthetic foot will then be replaced by a computerized prosthetic foot for one month, following which, the measurements will be repeated. Gait factors will be examined (spatio-temporal data, center of pressure movement) and internal loads inside the residuum will be evaluated. Comparison will also include patient's satisfaction and his ability to move around, evaluated by dedicated questionnaire.
  Interventions: Device: Elan foot prosthesis

INTERVENTIONS:
Device: Elan foot prosthesis — The research group will perform a gait analysis test (on a computerized treadmill) using their own non-computerized hydraulic foot, while in-socket pressures are measured. The prosthetic foot will then be replaced by a computerized prosthetic foot for one month, following which, the measurements will be repeated. Gait factors will be examined (spatio-temporal data, center of pressure movement) and internal loads inside the residuum will be evaluated. Comparison will also include patient's satisfaction and his ability to move around, evaluated by dedicated questionnaire.

SUMMARY:
Background:

Trauma is the second most common factor for transtibial amputations, just after vascular background. Traumatic amputees generally function better than amputees due to vascular background. The type of prosthetic foot fitted to the patient depends on his mobility and functional level, and significantly influences his stability and gait symmetry. A prosthetic foot with a hydraulic ankle provides significant advantages for high level functioning amputees: decrease of loads in the residuum, improvement in symmetry and generally gait pattern that is closer to natural. The hydraulic prosthetic foot has recently been upgraded to include computerized control over the ankle movement, using input from an array of sensors inside the foot. Studies have demonstrated decrease in energy consumption and gait pattern that is more similar to healthy people. However, hydraulic feet with and without computer control have not been compared. Furthermore, the effects of a computerized foot on various important factors have not been investigated yet, e.g. loads in the residuum, the movement of the center of pressure and the patient's satisfaction.

Research objectives:

To compare between hydraulic prosthetic feet, with and without computerized control. The comparison will be made while walking on flat or inclined surfaces (positive or negative inclination). Differences in gait parameters, loads inside the residuum, center of mass movement and patient's satisfaction will be quantified.

Research hypothesis: Using a computerized prosthetic foot will provide better mobility performances: improved gait factors and center of pressure movement, decrease internal loads in the residuum and increase patient's satisfaction.

Research design:

Clinical controlled research with research group(amputees) and control group (healthy).

DETAILED DESCRIPTION:
The research group will perform a gait analysis test (on a computerized treadmill) using their own non-computerized hydraulic foot, while in-socket pressures are measured. The prosthetic foot will then be replaced by a computerized prosthetic foot for one month, following which, the measurements will be repeated. Gait factors will be examined (spatio-temporal data, center of pressure movement) and internal loads inside the residuum will be evaluated. Comparison will also include patient's satisfaction and his ability to move around, evaluated by dedicated questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20 to 70 years old
* Traumatic unilateral Transtibial Amputee
* Using Echelon foot prosthesis for at least 6 months
* K level 3 or 4

Exclusion Criteria:

* Injury of the sound limb that compromises the gait of the amputee.

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Center of pressure movement | 2 to 6 weeks

SECONDARY OUTCOMES:
Pressure on the skin and internal loads in the residuum (measured by a surface pressure mapping technology). | 2 to 6 weeks
Grade in questionnaire for prosthetic evaluation. | 2 to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Itzhak Siev-Ner, MD, Principal Investigator — Sheba Medical Center